CLINICAL TRIAL: NCT07370246
Title: Evaluating the Safety and Efficacy of the Carotid Artery Stenting System for Stenosis With High-risk Features for CEA: a Prospective, Multicenter, Single-group Target-value Study in China
Brief Title: CAS for Stenosis With High-risk Features for CEA
Acronym: HeartCare CAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Shanghai HeartCare Medical Technology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QX2025-015-01
Record Dates: First submitted 2025-12-26; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Carotid Artery Stenosis; Carotid Artery Stenting
Keywords: Carotid artery stenosis; Carotid artery stent
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carotid artery stent system (Experimental): Device: The carotid artery stent system, manufactured by Shanghai HeartCare Medical Technology Co., Ltd., is a self-expanding stent constructed from nitinol.
  Interventions: Device: Carotid artery stent system

INTERVENTIONS:
Device: Carotid artery stent system — The carotid artery stent system consists of a nitinol self-expanding stent and a 1.65mm (5F) delivery device. At the tip of the delivery device and the inner part of the distal outer tube, there is a guidewire channel. The proximal end of the guidewire channel stops at the guidewire exchange port. The design allows for the accommodation of a guidewire with a diameter of 0.014inch (0.36mm).

SUMMARY:
The purpose of this prospective, multicenter, single-group target-value study is to evaluate the safety and efficacy of the carotid artery stent system in patients with high-risk features for carotid endarterectomy. This trial is utilizing the carotid artery stent system provided by Shanghai HeartCare Medical Technology Co., Ltd. and will be conducted at approximately 10 interventional neurology centers in China.

DETAILED DESCRIPTION:
This trial is a prospective, multicenter, single-group target-value study to evaluate the safety and efficacy of the carotid artery stent system in patients with high-risk features for carotid endarterectomy. The primary outcome is a composite outcome that includes stroke or death within 30 days after enrollment or after a revascularization procedure for the qualifying lesion during the follow-up period or ischemic stroke in the territory of the qualifying artery between day 31 and the end of the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, male or female;
2. Pre-procedural carotid duplex ultrasound and/or computed tomography angiography confirmed stenosis of the common carotid artery, internal carotid artery, or carotid bifurcation, and are considered suitable for endovascular treatment;
3. Intra-procedural digital subtraction angiography, using NASCET criteria, confirmed stenosis of ≥ 50% (symptomatic) or ≥ 80% (asymptomatic), and symptomatic is defined as the occurrence of one or more clinical events within 6 months prior to the procedure, including transient ischemic attack, amaurosis fugax, or minor/non-disabling stroke attributable to the ipsilateral intracranial circulation;
4. The vessel diameter of the target lesion is between 3.0 mm and 9.0 mm;
5. Voluntary participation in this trial and provision of written informed consent.

Inclusion criteria for high-risk features for carotid endarterectomy:

Comorbidity factors:

1. Age ≥ 75 years at the time of enrollment;
2. Patients with congestive heart failure (New York Heart Association Class III/IV);
3. Patients with unstable angina pectoris;
4. Patients with severe chronic obstructive pulmonary disease, defined as an FEV1 ≤ 50% of predicted, requirement for chronic oxygen therapy, or a resting PO₂ ≤ 60 mmHg;
5. Patients with left ventricular ejection fraction ≤ 30%;
6. Patients with recent myocardial infarction (within 2 to 6 weeks);
7. Patients with coronary artery disease with ≥ 70% stenosis in two or more major vessels;
8. Planned coronary artery bypass grafting or valve replacement surgery within 31 to 60 days following the procedure.

Anatomical factors:

1. Lesions located at or above the level of the second cervical vertebra (C2) or lesions that are surgically inaccessible below the clavicle;
2. History of radical head and neck surgery or radiotherapy;
3. Patients with limited cervical spine mobility;
4. Patients with tracheostomy;
5. History of vocal cord paralysis or laryngectomy;
6. Patients with contralateral recurrent laryngeal nerve palsy;
7. Patients with restenosis following previous carotid endarterectomy;
8. Patients with severe stenosis or occlusion of the contralateral carotid artery;
9. Severe tandem lesions that can be covered by a single stent.

Exclusion Criteria:

1. Target lesions caused by carotid arteritis;
2. Target lesions located at the origin of the common carotid artery;
3. Target lesions with extensive calcification or excessive tortuosity that preclude stent delivery;
4. Target lesions attributable to asymptomatic complete occlusion or the presence of a "string sign";
5. Target lesions adjacent to significant acute or subacute thrombus, or arteriovenous malformation;
6. History of major surgery (including intra-abdominal, intrathoracic, cardiac, or vascular procedures) within 30 days before the procedure, or any such surgery scheduled within 30 days after the procedure;
7. History of intracranial hemorrhage or progressive stroke within 3 months before the procedure;
8. History of an extensive hemispheric stroke within 2 weeks before the procedure;
9. History of bradycardia (heart rate < 40 bpm) before the procedure;
10. History of paroxysmal atrial fibrillation within the past 6 months, or paroxysmal atrial fibrillation requiring long-term anticoagulation therapy;
11. Patients with known or potential sources of thromboembolism (including previously known symptomatic patent foramen ovale, mechanical heart valves, or deep vein thrombosis treated within 6 months);
12. Patients with a known intracranial aneurysm requiring surgical intervention that cannot be treated before the procedure;
13. Patients with known coagulation disorders (APTT > 3 times the upper limit of normal) or abnormal bleeding disorders;
14. Patients with known contraindications to heparin or antiplatelet agents;
15. Patients with a platelet count < 100×10^9/L;
16. Patients with known allergies to any components of the investigational product, contrast agents;
17. Patients with known severe hepatic or renal insufficiency (ALT or AST > 5 times the upper limit of normal, or serum creatinine > 3 times the upper limit of normal);
18. Patients with known uncontrolled severe hypertension (persistent systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg);
19. Patients with a pre-procedure mRS score > 3;
20. Patients with extensively metastatic malignancy;
21. Patients concurrently enrolled in another drug or medical device clinical trial;
22. Female patients who are currently pregnant or breastfeeding, or who plan to conceive within 1 year;
23. Lesions inaccessible by endovascular approach (including severe tortuosity of aortic arch branches with no suitable access artery, or special aortic arch anatomy);
24. According to the judgment of the investigator, patients with an expected survival of less than 12 months;
25. According to the judgment of the investigator, other situations that are not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Stroke, myocardial infarction, and death within 30 days after the procedure, or stroke in the territory of the ipsilateral artery between day 31 and day 365 after the procedure | 30 days after the procedure and 365 days after the procedure
  Stroke is defined as an event that causes focal neurological dysfunction or signs and lasts for at least 24 hours, including ischemic stroke and hemorrhagic stroke. Myocardial infarction is defined as an increase in creatine kinase isoenzyme (CK-MB) or troponin in the postoperative period that is at least twice the upper limit of the normal range, accompanied by ischemic symptoms such as chest pain, or the presence of ischemic electrocardiogram evidence. Ischemic stroke in the territory of the ipsilateral artery is defined as an ischemic stroke in the cerebral hemisphere that is supplied with blood flow by the target artery.

SECONDARY OUTCOMES:
In-stent restenosis rate within 12 months after the procedure | 365 days after the procedure
  Angiography demonstrated restenosis of the target artery both within the 5-mm stent segment and at the stent margins, with a degree of stenosis ≥50%.
Implantation success rate | During the procedure
  Implantation success was defined as successful implantation of the stent (including delivery, release, and expansion), covering the target lesion area, and subsequent withdrawal of the delivery system.
Procedure success rate | Before the discharge or 7 days after the procedure
  Procedure success is defined as successful stent implantation followed by angiographic confirmation of ≤30% residual stenosis at the target lesion and the absence of any major adverse event prior to hospital discharge.
In-stent restenosis rate within 6 months after the procedure | 6 months after the procedure
  Angiography demonstrated restenosis of the target artery both within the 5-mm stent segment and at the stent margins, with a degree of stenosis ≥50%.
Symptomatic in-stent restenosis rate | 6 months, and 12 months after the procedure
  Symptomatic in-stent restenosis is defined as in-stent restenosis that results in an ischemic stroke or transient ischemic attack in the territory of the target artery.
Target lesion revascularization rate | 30 days, 6 months, and 12 months after the procedure
  Target lesion revascularization is defined as any repeat revascularization procedure performed on the original treatment site, encompassing the initial lesion segment and a 5-mm border zone proximal and distal to it.
Ischemic stroke in the territory of the ipsilateral artery between day 31 and day 365 after the procedure | 12 months after the procedure
  Ischemic stroke is defined as a new focal neurological deficit of sudden onset that is associated with an infarction lesion on CT or MRI.

OTHER OUTCOMES:
Major adverse event rate | 30 days, 6 months, 12 months after the procedure
  Major adverse events are defined as all deaths, strokes, and myocardial infarctions.
Adverse events rate | 30 days, 6 months, and 12 months after the procedure
Serious adverse events rate | 30 days, 6 months, and 12 months after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ning Ma, Professor, Principal Investigator — Beijing Tiantan Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yang B, Ma Y, Wang T, Chen Y, Wang Y, Zhao Z, Chen D, Wang J, Xu X, Luo T, Hua Y, Ling F, Qureshi AI, Hong B, Jiao L; RECAS Trial Investigators. Carotid Endarterectomy and Stenting in a Chinese Population: Safety Outcome of the Revascularization of Extracranial Carotid Artery Stenosis Trial. Transl Stroke Res. 2021 Apr;12(2):239-247. doi: 10.1007/s12975-020-00835-8. Epub 2020 Jul 19. PMID 32686047
- [Result] Ronchey S, Praquin B, Orrico M, Serrao E, Ciceroni C, Alberti V, Fazzini S, Mangialardi N. Outcomes of 1000 Carotid Wallstent Implantations: Single-Center Experience. J Endovasc Ther. 2016 Apr;23(2):267-74. doi: 10.1177/1526602815626558. Epub 2016 Jan 23. PMID 26802612
- [Result] Hopkins LN, White CJ, Foster MT, Powell RJ, Zemel G, Diaz-Cartelle J. Carotid artery stenting and patient outcomes: the CABANA surveillance study. Catheter Cardiovasc Interv. 2014 Nov 15;84(6):997-1004. doi: 10.1002/ccd.25578. Epub 2014 Jul 18. PMID 24948033
- [Result] Iyer SS, White CJ, Hopkins LN, Katzen BT, Safian R, Wholey MH, Gray WA, Ciocca R, Bachinsky WB, Ansel G, Joye JD, Russell ME; BEACH Investigators. Carotid artery revascularization in high-surgical-risk patients using the Carotid WALLSTENT and FilterWire EX/EZ: 1-year outcomes in the BEACH Pivotal Group. J Am Coll Cardiol. 2008 Jan 29;51(4):427-34. doi: 10.1016/j.jacc.2007.09.045. PMID 18222352
- [Result] White CJ, Iyer SS, Hopkins LN, Katzen BT, Russell ME; BEACH Trial Investigators. Carotid stenting with distal protection in high surgical risk patients: the BEACH trial 30 day results. Catheter Cardiovasc Interv. 2006 Apr;67(4):503-12. doi: 10.1002/ccd.20689. PMID 16548004
- [Result] Naylor R, Rantner B, Ancetti S, de Borst GJ, De Carlo M, Halliday A, Kakkos SK, Markus HS, McCabe DJH, Sillesen H, van den Berg JC, Vega de Ceniga M, Venermo MA, Vermassen FEG, Esvs Guidelines Committee, Antoniou GA, Bastos Goncalves F, Bjorck M, Chakfe N, Coscas R, Dias NV, Dick F, Hinchliffe RJ, Kolh P, Koncar IB, Lindholt JS, Mees BME, Resch TA, Trimarchi S, Tulamo R, Twine CP, Wanhainen A, Document Reviewers, Bellmunt-Montoya S, Bulbulia R, Darling RC 3rd, Eckstein HH, Giannoukas A, Koelemay MJW, Lindstrom D, Schermerhorn M, Stone DH. Editor's Choice - European Society for Vascular Surgery (ESVS) 2023 Clinical Practice Guidelines on the Management of Atherosclerotic Carotid and Vertebral Artery Disease. Eur J Vasc Endovasc Surg. 2023 Jan;65(1):7-111. doi: 10.1016/j.ejvs.2022.04.011. Epub 2022 May 20. No abstract available. PMID 35598721